CLINICAL TRIAL: NCT00818818
Title: Low-dose Pentavalent Antimony Treatment of Cutaneous Leishmaniasis in Old Age Patients Infected With Leishmania (Viannia) Braziliensis in Bahia State, Brazil. An Open Uncontrolled Trial.
Brief Title: Low-dose Pentavalent Antimony Treatment of Cutaneous Leishmaniasis in Old Age Patients
Acronym: Sbold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Brasilia (Other)
Responsible Party: Gustavo Adolfo Sierra Romero, Faculty of Medicine, University of Brasilia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lowdoseaging
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Localized Cutaneous Leishmaniasis
Keywords: Leishmaniasis; Cutaneous leishmaniasis; Leishmania braziliensis; Pentavalent antimonial; Glucantime
MeSH Terms: conditions — Leishmaniasis; Leishmaniasis, Cutaneous | interventions — Meglumine Antimoniate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meglumine antimoniate (Experimental): Treated with 5mg/kg/d of pentavalent antimony (meglumine antimoniate) intravenously for 20 consecutive days.
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Meglumine antimoniate — 5mg/kg/d of pentavalent antimony, IV, for 20 consecutive days
  Other Names: Glucantime

SUMMARY:
This study was designed to evaluate the effect of low doses of pentavalent antimony (meglumine antimoniate) to treat cutaneous leishmaniasis ulcers in patients older than 65 years. The hypothesis is that older patients may have a positive response with a lower dose of pentavalent antimony, avoiding the frequent adverse events observed with the standard dose. The design is that of an open uncontrolled trial enrolling 20 patients infected with the parasite Leishmania braziliensis in an endemic area of the State of Bahia, Brazil. The endpoint of cure or therapeutic failure will be evaluated at the third month of follow-up after treatment to avoid the impact of spontaneous cure as a confounding factor.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Permanent residence in the endemic area
* Availability of a caregiver for dependent patients

Exclusion Criteria:

* Mucosal disease caused by leishmaniasis
* Disseminated cutaneous disease
* Severe cardiac, renal or hepatic disorders
* Active cancer
* Active tuberculosis
* Leprosy
* HIV positive
* Total bilirubin > 1.5mg/dL
* Urea and creatinin > 1.5 times the upper normal level
* Alkaline phosphatase and aminotransferases > 2.5 times the upper normal level
* Lipase and amylase > 1.5 the upper normal level
* Hemoglobin < 5 g/dL of

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Clinical cure | Three months after treatment
  Clinical cure defined as the complete epithelialization of the ulcerated lesions without any inflamatory sign (erythema, edema, disquamation)

SECONDARY OUTCOMES:
Adverse events rate - day 7 | 7th day
  Biochemical abnormalities detected in serum samples for: SGOT, SGPT, amilase, creatinin, ureia and glycemia, or any sign or symptom experienced during the first week of treatment
Adverse events rate - day 14 | 14th day
  Biochemical abnormalities detected in serum samples for: SGOT, SGPT, amilase, creatinin, ureia and glycemia, or any sign or symptom experienced during the second week of treatment
Total Adverse events rate | 20th day
  Biochemical abnormalities detected in serum samples for: SGOT, SGPT, amilase, creatinin, ureia and glycemia, or any sign or symptom experienced during the whole treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julia S Ampuero-Vela, MD, MSc, Principal Investigator — Faculty of Medicine, University of Brasilia; Gustavo Adolfo S Romero, MD, PhD, Study Chair — Faculty of Medicine, University of Brasilia
Locations (1):
- Health Center Unit of Corte de Pedra, Corte de Pedra, Presidente Tancredo Neves, Bahia State, Brazil